CLINICAL TRIAL: NCT01314313
Title: Edwards SAPIEN XT Transcatheter Heart Valve Therapy for Intermediate and High Risk Patients
Brief Title: PARTNER II Trial: Placement of AoRTic TraNscathetER Valves II - XT Intermediate and High Risk
Acronym: PII A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12 PIIA
Record Dates: First submitted 2011-03-07; First posted 2011-03-14 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: SAPIEN XT; Transfemoral; Transapical; Transaortic; NovaFlex; TAVI; Aortic Stenosis; THV; Aortic Valve; Transcatheter Heart Valve; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PIIA - SAPIEN XT (Experimental): PIIA is operable group
  Interventions: Device: TAVR Implantation with SAPIEN XT
- Control: SAVR (Active Comparator): SAVR (surgical aortic valve replacement) is the control arm
  Interventions: Device: SAVR Implantation

INTERVENTIONS:
Device: TAVR Implantation with SAPIEN XT — Operable Group with SAPIEN XT
  Arms: PIIA - SAPIEN XT
Device: SAVR Implantation — Control Group
  Arms: Control: SAVR

SUMMARY:
The purpose of this trial is to determine the safety and effectiveness of the Edwards SAPIEN XT transcatheter heart valve and delivery systems which are intended for use in patients with symptomatic, calcific, severe aortic stenosis.

DETAILED DESCRIPTION:
The PIIA cohort is a prospective multi-center trial undergoing aortic valve replacement for severe aortic stenosis. Patients randomized to the treatment arm will receive an Edwards SAPIEN XT THV with either transfemoral, transapical or transaortic delivery access. Patients in the control arm will receive a surgical bioprosthetic heart valve via aortic valve replacement surgery.

To assure that patients with an STS score ≥ 4% have been selected.

ELIGIBILITY:
Inclusion Criteria

1. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s and an initial aortic valve area (AVA) of ≤0.8 cm2 or indexed EOA < 0.5 cm2/m2 Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
3. The heart team agrees (and verified in the case review process) that valve implantation will likely benefit the patient.
4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which will be conducted as a phone follow-up.
6. Study patient agrees to undergo surgical aortic valve replacement (SAVR) - if randomized to control treatment.

Exclusion Criteria

1. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
2. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified.
3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
4. Preexisting mechanical or bioprosthetic valve in any position (except NR3).
5. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker or ICD (S3 Cohort only) is not excluded.
6. Heart team assessment of inoperability (including examining cardiac surgeon).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2032 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University; Craig Smith, MD, Principal Investigator — Columbia University
Locations (57):
- United States (55):
  - Arkansas Heart Hospital/Clinic, Little Rock, Arkansas
  - Scripps Green Hospital, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Miami Hospital Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Northshore, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - The University of Iowa, Iowa City, Iowa
  - The Jewish Hospital Medical Center, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic-Saint Marys Hospital, Rochester, Minnesota
  - St. Luke's Hospital - Mid America Heart Institute, Kansas City, Missouri
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University, Camden, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - New York Presbyterian Hospital - Cornell, New York, New York
  - Columbia University Medical Center, New York, New York
  - East Carolina Heart Institute at East Carolina University, Greenville, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute at Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Austin Heart, PLLC, Austin, Texas
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - Medical City Dallas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio (UTHSCSA), San Antonio, Texas
  - IHC Health Services Inc. dba Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (2):
  - St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhavan MV, Kodali SK, Thourani VH, Makkar R, Mack MJ, Kapadia S, Webb JG, Cohen DJ, Herrmann HC, Williams M, Greason K, Pibarot P, Hahn RT, Jaber W, Xu K, Alu M, Smith CR, Leon MB. Outcomes of SAPIEN 3 Transcatheter Aortic Valve Replacement Compared With Surgical Valve Replacement in Intermediate-Risk Patients. J Am Coll Cardiol. 2023 Jul 11;82(2):109-123. doi: 10.1016/j.jacc.2023.04.049. PMID 37407110
- [Derived] Genereux P, Pibarot P, Redfors B, Bax JJ, Zhao Y, Makkar RR, Kapadia S, Thourani VH, Mack MJ, Nazif TM, Lindman BR, Babaliaros V, Vincent F, Russo M, McCabe JM, Gillam LD, Alu MC, Hahn RT, Webb JG, Leon MB, Cohen DJ. Evolution and Prognostic Impact of Cardiac Damage After Aortic Valve Replacement. J Am Coll Cardiol. 2022 Aug 23;80(8):783-800. doi: 10.1016/j.jacc.2022.05.006. Epub 2022 May 17. PMID 35595203
- [Derived] Vincent F, Thourani VH, Ternacle J, Redfors B, Cohen DJ, Hahn RT, Li D, Crowley A, Webb JG, Mack MJ, Kapadia S, Russo M, Smith CR, Alu MC, Leon MB, Pibarot P. Time-of-Day and Clinical Outcomes After Surgical or Transcatheter Aortic Valve Replacement: Insights From the PARTNER Trials. Circ Cardiovasc Qual Outcomes. 2022 Jan;15(1):e007948. doi: 10.1161/CIRCOUTCOMES.121.007948. Epub 2022 Jan 18. PMID 35041482
- [Derived] Abbas AE, Ternacle J, Pibarot P, Xu K, Alu M, Rogers E, Hahn RT, Leon M, Thourani VH. Impact of Flow on Prosthesis-Patient Mismatch Following Transcatheter and Surgical Aortic Valve Replacement. Circ Cardiovasc Imaging. 2021 Aug;14(8):e012364. doi: 10.1161/CIRCIMAGING.120.012364. Epub 2021 Aug 13. PMID 34387097
- [Derived] Cremer PC, Wang TKM, Rodriguez LL, Lindman BR, Zhang Y, Zajarias A, Hahn RT, Lerakis S, Malaisrie SC, Douglas PS, Pibarot P, Svensson LG, Kapadia S, Leon MB, Jaber WA; PARTNER II Investigators. Incidence and Clinical Significance of Worsening Tricuspid Regurgitation Following Surgical or Transcatheter Aortic Valve Replacement: Analysis From the PARTNER IIA Trial. Circ Cardiovasc Interv. 2021 Aug;14(8):e010437. doi: 10.1161/CIRCINTERVENTIONS.120.010437. Epub 2021 Jul 16. PMID 34266311
- [Derived] Brener MI, George I, Kosmidou I, Nazif T, Zhang Z, Dizon JM, Garan H, Malaisrie SC, Makkar R, Mack M, Szeto WY, Fearon WF, Thourani VH, Leon MB, Kodali S, Biviano AB. Atrial Fibrillation Is Associated With Mortality in Intermediate Surgical Risk Patients With Severe Aortic Stenosis: Analyses From the PARTNER 2A and PARTNER S3i Trials. J Am Heart Assoc. 2021 Apr 6;10(7):e019584. doi: 10.1161/JAHA.120.019584. Epub 2021 Mar 23. PMID 33754803
- [Derived] Pibarot P, Ternacle J, Jaber WA, Salaun E, Dahou A, Asch FM, Weissman NJ, Rodriguez L, Xu K, Annabi MS, Guzzetti E, Beaudoin J, Bernier M, Leipsic J, Blanke P, Clavel MA, Rogers E, Alu MC, Douglas PS, Makkar R, Miller DC, Kapadia SR, Mack MJ, Webb JG, Kodali SK, Smith CR, Herrmann HC, Thourani VH, Leon MB, Hahn RT; PARTNER 2 Investigators. Structural Deterioration of Transcatheter Versus Surgical Aortic Valve Bioprostheses in the PARTNER-2 Trial. J Am Coll Cardiol. 2020 Oct 20;76(16):1830-1843. doi: 10.1016/j.jacc.2020.08.049. PMID 33059828
- [Derived] Makkar RR, Thourani VH, Mack MJ, Kodali SK, Kapadia S, Webb JG, Yoon SH, Trento A, Svensson LG, Herrmann HC, Szeto WY, Miller DC, Satler L, Cohen DJ, Dewey TM, Babaliaros V, Williams MR, Kereiakes DJ, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Brown DL, Fearon WF, Russo MJ, Pibarot P, Hahn RT, Jaber WA, Rogers E, Xu K, Wheeler J, Alu MC, Smith CR, Leon MB; PARTNER 2 Investigators. Five-Year Outcomes of Transcatheter or Surgical Aortic-Valve Replacement. N Engl J Med. 2020 Jan 29;382(9):799-809. doi: 10.1056/NEJMoa1910555. Print 2020 Feb 27. PMID 31995682
- [Derived] Chen S, Redfors B, O'Neill BP, Clavel MA, Pibarot P, Elmariah S, Nazif T, Crowley A, Ben-Yehuda O, Finn MT, Alu MC, Vahl TP, Kodali S, Leon MB, Lindman BR. Low and elevated B-type natriuretic peptide levels are associated with increased mortality in patients with preserved ejection fraction undergoing transcatheter aortic valve replacement: an analysis of the PARTNER II trial and registry. Eur Heart J. 2020 Feb 21;41(8):958-969. doi: 10.1093/eurheartj/ehz892. PMID 31883339
- [Derived] Summers MR, Leon MB, Smith CR, Kodali SK, Thourani VH, Herrmann HC, Makkar RR, Pibarot P, Webb JG, Leipsic J, Alu MC, Crowley A, Hahn RT, Kapadia SR, Tuzcu EM, Svensson L, Cremer PC, Jaber WA. Prosthetic Valve Endocarditis After TAVR and SAVR: Insights From the PARTNER Trials. Circulation. 2019 Dec 10;140(24):1984-1994. doi: 10.1161/CIRCULATIONAHA.119.041399. Epub 2019 Nov 6. PMID 31690104
- [Derived] Furer A, Chen S, Redfors B, Elmariah S, Pibarot P, Herrmann HC, Hahn RT, Kodali S, Thourani VH, Douglas PS, Alu MC, Fearon WF, Passeri J, Malaisrie SC, Crowley A, McAndrew T, Genereux P, Ben-Yehuda O, Leon MB, Burkhoff D. Effect of Baseline Left Ventricular Ejection Fraction on 2-Year Outcomes After Transcatheter Aortic Valve Replacement: Analysis of the PARTNER 2 Trials. Circ Heart Fail. 2019 Aug;12(8):e005809. doi: 10.1161/CIRCHEARTFAILURE.118.005809. Epub 2019 Aug 1. PMID 31525069
- [Derived] Nazif TM, Chen S, George I, Dizon JM, Hahn RT, Crowley A, Alu MC, Babaliaros V, Thourani VH, Herrmann HC, Smalling RW, Brown DL, Mack MJ, Kapadia S, Makkar R, Webb JG, Leon MB, Kodali SK. New-onset left bundle branch block after transcatheter aortic valve replacement is associated with adverse long-term clinical outcomes in intermediate-risk patients: an analysis from the PARTNER II trial. Eur Heart J. 2019 Jul 14;40(27):2218-2227. doi: 10.1093/eurheartj/ehz227. PMID 31505615
- [Derived] Chakravarty T, Patel A, Kapadia S, Raschpichler M, Smalling RW, Szeto WY, Abramowitz Y, Cheng W, Douglas PS, Hahn RT, Herrmann HC, Kereiakes D, Svensson L, Yoon SH, Babaliaros VC, Kodali S, Thourani VH, Alu MC, Liu Y, McAndrew T, Mack M, Leon MB, Makkar RR. Anticoagulation After Surgical or Transcatheter Bioprosthetic Aortic Valve Replacement. J Am Coll Cardiol. 2019 Sep 3;74(9):1190-1200. doi: 10.1016/j.jacc.2019.06.058. PMID 31466616
- [Derived] Baron SJ, Wang K, House JA, Magnuson EA, Reynolds MR, Makkar R, Herrmann HC, Kodali S, Thourani VH, Kapadia S, Svensson L, Mack MJ, Brown DL, Russo MJ, Smith CR, Webb J, Miller C, Leon MB, Cohen DJ. Cost-Effectiveness of Transcatheter Versus Surgical Aortic Valve Replacement in Patients With Severe Aortic Stenosis at Intermediate Risk. Circulation. 2019 Feb 12;139(7):877-888. doi: 10.1161/CIRCULATIONAHA.118.035236. PMID 30586747
- [Derived] Pibarot P, Hahn RT, Weissman NJ, Arsenault M, Beaudoin J, Bernier M, Dahou A, Khalique OK, Asch FM, Toubal O, Leipsic J, Blanke P, Zhang F, Parvataneni R, Alu M, Herrmann H, Makkar R, Mack M, Smalling R, Leon M, Thourani VH, Kodali S. Association of Paravalvular Regurgitation With 1-Year Outcomes After Transcatheter Aortic Valve Replacement With the SAPIEN 3 Valve. JAMA Cardiol. 2017 Nov 1;2(11):1208-1216. doi: 10.1001/jamacardio.2017.3425. PMID 28973091
- [Derived] Baron SJ, Arnold SV, Wang K, Magnuson EA, Chinnakondepali K, Makkar R, Herrmann HC, Kodali S, Thourani VH, Kapadia S, Svensson L, Brown DL, Mack MJ, Smith CR, Leon MB, Cohen DJ; PARTNER 2 Investigators. Health Status Benefits of Transcatheter vs Surgical Aortic Valve Replacement in Patients With Severe Aortic Stenosis at Intermediate Surgical Risk: Results From the PARTNER 2 Randomized Clinical Trial. JAMA Cardiol. 2017 Aug 1;2(8):837-845. doi: 10.1001/jamacardio.2017.2039. PMID 28658491
- [Derived] Webb JG, Mack MJ, White JM, Dvir D, Blanke P, Herrmann HC, Leipsic J, Kodali SK, Makkar R, Miller DC, Pibarot P, Pichard A, Satler LF, Svensson L, Alu MC, Suri RM, Leon MB. Transcatheter Aortic Valve Implantation Within Degenerated Aortic Surgical Bioprostheses: PARTNER 2 Valve-in-Valve Registry. J Am Coll Cardiol. 2017 May 9;69(18):2253-2262. doi: 10.1016/j.jacc.2017.02.057. PMID 28473128
- [Derived] Blanke P, Pibarot P, Hahn R, Weissman N, Kodali S, Thourani V, Parvataneni R, Dvir D, Naoum C, Norgaard BL, Douglas P, Jaber W, Khalique OK, Jilaihawi H, Mack M, Smith C, Leon M, Webb J, Leipsic J. Computed Tomography-Based Oversizing Degrees and Incidence of Paravalvular Regurgitation of a New Generation Transcatheter Heart Valve. JACC Cardiovasc Interv. 2017 Apr 24;10(8):810-820. doi: 10.1016/j.jcin.2017.02.021. PMID 28427598
- [Derived] Herrmann HC, Thourani VH, Kodali SK, Makkar RR, Szeto WY, Anwaruddin S, Desai N, Lim S, Malaisrie SC, Kereiakes DJ, Ramee S, Greason KL, Kapadia S, Babaliaros V, Hahn RT, Pibarot P, Weissman NJ, Leipsic J, Whisenant BK, Webb JG, Mack MJ, Leon MB; PARTNER Investigators. One-Year Clinical Outcomes With SAPIEN 3 Transcatheter Aortic Valve Replacement in High-Risk and Inoperable Patients With Severe Aortic Stenosis. Circulation. 2016 Jul 12;134(2):130-40. doi: 10.1161/CIRCULATIONAHA.116.022797. PMID 27400898
- [Derived] Kodali S, Thourani VH, White J, Malaisrie SC, Lim S, Greason KL, Williams M, Guerrero M, Eisenhauer AC, Kapadia S, Kereiakes DJ, Herrmann HC, Babaliaros V, Szeto WY, Hahn RT, Pibarot P, Weissman NJ, Leipsic J, Blanke P, Whisenant BK, Suri RM, Makkar RR, Ayele GM, Svensson LG, Webb JG, Mack MJ, Smith CR, Leon MB. Early clinical and echocardiographic outcomes after SAPIEN 3 transcatheter aortic valve replacement in inoperable, high-risk and intermediate-risk patients with aortic stenosis. Eur Heart J. 2016 Jul 21;37(28):2252-62. doi: 10.1093/eurheartj/ehw112. Epub 2016 Mar 31. PMID 27190101
- [Derived] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Derived] Webb JG, Doshi D, Mack MJ, Makkar R, Smith CR, Pichard AD, Kodali S, Kapadia S, Miller DC, Babaliaros V, Thourani V, Herrmann HC, Bodenhamer M, Whisenant BK, Ramee S, Maniar H Jr, Kereiakes D, Xu K, Jaber WA, Menon V, Tuzcu EM, Wood D, Svensson LG, Leon MB. A Randomized Evaluation of the SAPIEN XT Transcatheter Heart Valve System in Patients With Aortic Stenosis Who Are Not Candidates for Surgery. JACC Cardiovasc Interv. 2015 Dec 21;8(14):1797-806. doi: 10.1016/j.jcin.2015.08.017. PMID 26718510
- [Derived] Haussig S, Linke A. Patient selection for TAVI 2015 - TAVI in low-risk patients: fact or fiction? EuroIntervention. 2015 Sep;11 Suppl W:W86-91. doi: 10.4244/EIJV11SWA27. PMID 26384204
- [Derived] Lindman BR, Maniar HS, Jaber WA, Lerakis S, Mack MJ, Suri RM, Thourani VH, Babaliaros V, Kereiakes DJ, Whisenant B, Miller DC, Tuzcu EM, Svensson LG, Xu K, Doshi D, Leon MB, Zajarias A. Effect of tricuspid regurgitation and the right heart on survival after transcatheter aortic valve replacement: insights from the Placement of Aortic Transcatheter Valves II inoperable cohort. Circ Cardiovasc Interv. 2015 Apr;8(4):10.1161/CIRCINTERVENTIONS.114.002073 e002073. doi: 10.1161/CIRCINTERVENTIONS.114.002073. PMID 25855679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 23, 2011 to November 6, 2013 2,032 patients were enrolled into the PARTNER II A SAPIEN XT vs SAVR Intermediate Risk Trial at 57 sites in the United States and Canada.
Groups:
- PIIA: SAPIEN XT: Edwards SAPIEN XT Transcatheter Heart Valve (THV)
  NOTE: SAVR with surgical bioprosthetic heart valve is the control arm.
- Control: SAVR: Surgical Aortic Valve Replacement (SAVR)
Period: Overall Study
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Started | 1011 | 1021
As Treated | 994 | 944
Valve Implanted | 974 | 936
Completed (This is two year follow-up) | 784 | 710
Not Completed | 227 | 311

BASELINE CHARACTERISTICS:
Groups:
- PIIA: SAPIEN XT: Edwards SAPIEN XT Transcatheter Heart Valve (THV)
- Control: SAVR: Surgical Aortic Valve Replacement (SAVR); Control for PIIA: SAPIEN XT
- Total: Total of all reporting groups
Arm/Group | PIIA: SAPIEN XT | Control: SAVR | Total
Number analyzed (Participants) | 1011 | 1021 | 2032
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.5 (6.70) | 81.7 (6.71) | 81.6 (6.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 463 | 461 | 924
  Male | 548 | 560 | 1108
STS Score [Mean (Standard Deviation); unit: % risk of mortality or morbidity] — The Society of Thoracic Surgeons (STS) score measures patient risk at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  % risk of mortality or morbidity | 5.8 (2.08) | 5.8 (1.87) | 5.8 (1.98)
NYHA Classification [Number; unit: participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  participants
    NYHA I/II | 229 | 244 | 473
    NYHA III/VI | 782 | 776 | 1558

OUTCOME MEASURES:

1. Primary Outcome: All-cause Death or Disabling Stroke to Two Years
Description: All-cause Death or Disabling Stroke (Edwards SAPIEN XT THV vs SAVR)
Time Frame: 2 Years
Population: Participants include all patients who were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Control: SAVR: Control: Surgical Aortic Valve Replacement (SAVR)
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 1011 | 1021
Participants | 192 | 202

2. Secondary Outcome: Adjusted Days Alive and Out of Hospital (DAOH) to Two Years
Description: The number of days the patients are alive and out of the hospital.
Time Frame: 2 years
Population: Intent to Treat Population: All randomized patients with the exception of Total Aortic Regurgitation and Effective Orifice Area which was analyzed with the Valve Implant Population: All randomized patients receiving the valve.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 998 | 953
days | 629.4 (208.54) | 597.8 (236.80)

3. Secondary Outcome: Total Aortic Regurgitation (AR) at 2 Years
Description: Total aortic regurgitation was assessed by the core lab as "Grade 0" = None, "Grade 1+" = Trace, "Grade 2+" = Mild, "Grade 3+" = Moderate and "Grade 4+" = Severe. Total regurgitation at two year was analyzed in the valve implant population.
Time Frame: 2 years
Population: All randomized patients who received the valve were analyzed. Note: Echos were not available for all the patients who made the follow-up visit.
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 606 | 520
Grade | 1.2 (1.0) | 0.5 (0.7)

4. Secondary Outcome: 6MWT Change From Baseline
Description: Six Minute Walk Test change from baseline to 2 years
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 604 | 1021
meters | 14.5 (128.7) | NA (NA) — This secondary endpoint analyzes change within the SAPIEN XT Cohort.

5. Secondary Outcome: NYHA Classification at 2 Years
Description: New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PIIA: SAPIEN XT: Intermediate Risk Surgical Patients: Transcatheter Heart Valve (THV)
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 737 | 649
units on a scale | 1.5 (0.7) | 1.4 (0.6)

6. Secondary Outcome: Effective Orifice Area (EOA)
Time Frame: 2 years
Population: Effective Orifice Area is listed for only the patients who had echo available at the follow-up visit.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | PIIA: SAPIEN XT | Control: SAVR
Number analyzed (Participants) | 573 | 490
cm^2 | 1.5 (0.4) | 1.4 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse event data are currently available and reported for all events at 2 years were reported at the time of database lock.
Description: Adverse Events are site reported. Only Valve-Implanted patients are reported for all adverse events (except for mortality).
Groups:
- PIIA: SAPIEN XT - 2 Year: Edwards SAPIEN XT Transcatheter Heart Valve (THV)
- Control: SAVR - 2 Year: Surgical Aortic Valve Replacement (SAVR)
  NOTE: SAVR with surgical bioprosthetic heart valve is the control arm.
Arm/Group | PIIA: SAPIEN XT - 2 Year | Control: SAVR - 2 Year
All-Cause Mortality (participants affected / at risk) | 166/1011 | 170/1021
Serious Adverse Events (participants affected / at risk) | 666/974 | 672/936
Other Adverse Events (participants affected / at risk) | 838/974 | 864/936
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIIA: SAPIEN XT - 2 Year (N=974) | Control: SAVR - 2 Year (N=936)
Abnormal lab value (Investigations) | 24 (28) | 42 (46)
Access site and access related vascular injury - Aortic root rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Access site and access related vascular injury - Dissection (Injury, poisoning and procedural complications) | 20 (21) | 8 (8)
Access site/access related vascular injury - Distal embolization (noncerebral) from vascular source (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Access site/related vascular injury - Failure of perc access site closure causing intervention (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Access site and access related vascular injury - Hematoma (Injury, poisoning and procedural complications) | 2 (3) | 5 (5)
Access site and access related vascular injury - Perforation (Injury, poisoning and procedural complications) | 9 (9) | 7 (7)
Access site and access related vascular injury - Pseudoaneurysm (Injury, poisoning and procedural complications) | 10 (10) | 1 (1)
Access site and access related vascular injury - Rupture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Access site and access related vascular injury - Stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Access site and access related vascular injury - Ventricular rupture (Apical rupture) (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 24 (26) | 38 (43)
Anesthesia related complication - Aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anesthesia related complication - Confusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anesthesia related complication - Dysphasia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anesthesia related complication - Other (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Angina/Cardiac chest pain (Cardiac disorders) | 22 (28) | 24 (30)
Aortic insufficiency/Regurgitation PV leak - Non structural dysfunction (General disorders) | 24 (30) | 8 (9)
Aortic insufficiency/Regurgitation PV leak - Structural dysfunction (General disorders) | 7 (7) | 1 (1)
Aortic insufficiency/Regurgitation non valvular cause (General disorders) | 2 (3) | 0 (0)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 170 (186) | 196 (226)
Bleeding - Hemorrhage (Vascular disorders) | 145 (167) | 248 (297)
Cardiac arrest (Cardiac disorders) | 33 (33) | 36 (38)
Cardiac tamponade/Pericardial effusion (Cardiac disorders) | 21 (21) | 13 (13)
Cardiogenic shock (Cardiac disorders) | 9 (9) | 20 (20)
Coronary flow obstruction/Transvalvular flow disturbance (General disorders) | 6 (9) | 8 (8)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2)
Device embolization (General disorders) | 6 (6) | 0 (0)
Device migration/malposition requiring intervention (General disorders) | 6 (6) | 0 (0)
Edema (General disorders) | 7 (7) | 7 (7)
Embolization including air/calcific valve material or Thrombus (Vascular disorders) | 15 (15) | 26 (27)
Encephalopathy (Nervous system disorders) | 7 (7) | 4 (4)
Exercise intolerance or weakness (General disorders) | 2 (2) | 2 (2)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 67 (77) | 53 (65)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 18 (18) | 10 (10)
Heart failure/CHF/Low output failure (Cardiac disorders) | 127 (197) | 103 (134)
Hypertension (Vascular disorders) | 6 (6) | 3 (3)
Hypotension (Vascular disorders) | 14 (14) | 24 (25)
Infection - Access site infection (Infections and infestations) | 16 (17) | 2 (2)
Infection - Bacteremia (Infections and infestations) | 14 (15) | 13 (14)
Infection - Endocarditis (Infections and infestations) | 14 (15) | 11 (11)
Infection - Other (Infections and infestations) | 37 (48) | 56 (67)
Infection - Respiratory infection (Infections and infestations) | 93 (110) | 100 (111)
Infection - Sepsis (Infections and infestations) | 41 (44) | 47 (52)
Infection - Sternal wound infection (Infections and infestations) | 1 (1) | 14 (18)
Infection - Urinary tract infection (Infections and infestations) | 40 (47) | 31 (36)
Ischemia (Vascular disorders) | 13 (20) | 21 (24)
MI (Cardiac disorders) | 29 (29) | 26 (30)
Mental state change (not neurological) - Confusion (Psychiatric disorders) | 14 (14) | 14 (16)
Mental state change (not neurological) - Dementia (Nervous system disorders) | 7 (8) | 4 (5)
Mental state change (not neurological) - Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Miscellaneous - Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (31) | 26 (28)
Miscellaneous - Drug reaction (General disorders) | 2 (2) | 6 (6)
Miscellaneous - Fall (Injury, poisoning and procedural complications) | 25 (26) | 32 (34)
Miscellaneous - Other (General disorders) | 22 (28) | 23 (24)
Miscellaneous - Suicide (General disorders) | 1 (1) | 0 (0)
Mitral valve injury or insufficiency (Cardiac disorders) | 1 (1) | 2 (2)
Multi organ failure (General disorders) | 4 (4) | 10 (10)
Musculoskeletal - Fracture (Musculoskeletal and connective tissue disorders) | 47 (51) | 43 (45)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 33 (35) | 32 (35)
Neurological - Change in level of consciousness (Nervous system disorders) | 0 (0) | 6 (6)
Neurological - Cognitive impairment (Psychiatric disorders) | 0 (0) | 3 (3)
Neurological - Dysphasia/Aphasia (Nervous system disorders) | 5 (6) | 0 (0)
Neurological - Hemianopia (blindness in one half of the visual field) (Nervous system disorders) | 0 (0) | 2 (2)
Neurological - Hemiparesis (One sided body weakness) (Nervous system disorders) | 1 (1) | 6 (6)
Neurological - Hemiplegia (One side limb weakness) (Nervous system disorders) | 0 (0) | 3 (3)
Neurological - Hemorrhagic stroke (Nervous system disorders) | 15 (15) | 11 (12)
Neurological - Ischemic stroke (Nervous system disorders) | 57 (58) | 46 (47)
Neurological - Other (Nervous system disorders) | 18 (20) | 24 (25)
Neurological - Other new neurological sign consistent with stroke (Nervous system disorders) | 6 (6) | 4 (4)
Neurological - Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Neurological - TIA (Nervous system disorders) | 22 (23) | 14 (15)
Neurological - Undetermined stroke (Nervous system disorders) | 9 (9) | 5 (5)
Other (General disorders) | 70 (80) | 68 (72)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2)
Renal insufficiency or renal failure (Renal and urinary disorders) | 48 (53) | 80 (88)
Respiratory event - Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (10)
Respiratory event - Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory event - Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 21 (24)
Respiratory event - Other (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 18 (19)
Respiratory event - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 16 (18)
Respiratory event - Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Respiratory event - Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 64 (81)
Respiratory event - Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 50 (56) | 75 (92)
Syncope (Vascular disorders) | 21 (22) | 20 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 24 (24)
Unknown cause of death (General disorders) | 21 (21) | 19 (19)
Valve stenosis - Restenosis (General disorders) | 1 (1) | 1 (1)
Valve thrombosis (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIIA: SAPIEN XT - 2 Year (N=974) | Control: SAVR - 2 Year (N=936)
Abnormal lab value (Investigations) | 187 (260) | 257 (404)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 168 (192) | 198 (219)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 284 (338) | 409 (507)
Bleeding - Hemorrhage (Vascular disorders) | 285 (345) | 421 (500)
Edema (General disorders) | 39 (40) | 53 (56)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 96 (108) | 125 (157)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 47 (54) | 58 (64)
Heart failure/CHF/Low output failure (Cardiac disorders) | 71 (75) | 90 (101)
Hypertension (Vascular disorders) | 74 (75) | 48 (49)
Hypotension (Vascular disorders) | 56 (62) | 97 (102)
Infection - Other (Infections and infestations) | 86 (96) | 84 (96)
Infection - Respiratory infection (Infections and infestations) | 98 (112) | 101 (118)
Infection - Urinary tract infection (Infections and infestations) | 133 (164) | 165 (198)
Mental state change (not neurological) - Confusion (Psychiatric disorders) | 39 (42) | 63 (65)
Miscellaneous - Fall (Injury, poisoning and procedural complications) | 80 (94) | 66 (76)
Miscellaneous - Other (General disorders) | 62 (72) | 67 (81)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 100 (121) | 90 (108)
Other (General disorders) | 165 (213) | 175 (221)
Renal insufficiency or renal failure (Renal and urinary disorders) | 214 (254) | 258 (297)
Respiratory event - Atelectasis (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 51 (51)
Respiratory event - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 47 (49)
Respiratory Event - Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 70 (75) | 178 (191)
Thrombocytopenia (Blood and lymphatic system disorders) | 120 (126) | 210 (217)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes